CLINICAL TRIAL: NCT00667862
Title: A Phase II, Open Label, Single Arm Study of i.v. Panobinostat (LBH589) in Patients With Metastatic Hormone Refractory Prostate Cancer
Brief Title: Efficacy and Safety Study of Panobinostat in Participants With Metastatic Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589C2208; 2007-004995-37 (EudraCT Number)
Record Dates: First submitted 2008-04-18; First posted 2008-04-28 (Estimated); Results first posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-05

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Adenocarcinoma; Prostate-Specific Antigen; metastatic; male; HRPC; DACi
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Adenocarcinoma; Neoplasm Metastasis | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Panobinostat (Experimental): Participants with metastatic hormone refractory prostate cancer received 20 milligrams per meter square (mg/m^2) of panobinostat intravenously (i.v.) on Days 1 and 8 of a 21-day cycle. Treatment continued until disease progression as per investigator, intolerable toxicity, start of new cancer therapy, death, or withdrawal of consent.
  Interventions: Drug: Panobinostat

INTERVENTIONS:
Drug: Panobinostat
  Other Names: LBH589

SUMMARY:
This Phase II single dose study was designed to characterize the safety, tolerability, and efficacy of intravenous (i.v.) panobinostat as a single-agent treatment in participants with hormone refractory prostate cancer.

ELIGIBILITY:
Inclusion criteria:

* Confirmed diagnosis of adenocarcinoma of the prostate
* Participants with metastatic hormone refractory prostate cancer
* Participants that have had at least one, but not more than two prior cytotoxic treatments for prostate cancer
* Evidence of disease progression by at least one of the following:

  1. two or more lesions on bone scan
  2. progressive measurable disease
  3. two documented increases in prostate-specific antigen (PSA)
* Willing to use contraception throughout the study and for 12 weeks after study completion

Exclusion criteria:

* History or clinical signs of central nervous system (CNS) disease
* History of other cancers not curatively treated with no evidence of disease for more than 5 years
* Prior radiotherapy within 3 weeks of starting study treatment
* Prior radiopharmaceuticals (strontium, samarium)
* Impaired cardiac function
* Heart disease
* Liver or renal disease with impaired function

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male participants are eligible as it is a prostate cancer study.
Enrollment: 35 (Actual)
Dates: Start 2008-03-18 (Actual); Primary Completion 2010-11-05 (Actual); Study Completion 2010-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (5):
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Background] Rathkopf DE, Picus J, Hussain A, Ellard S, Chi KN, Nydam T, Allen-Freda E, Mishra KK, Porro MG, Scher HI, Wilding G. A phase 2 study of intravenous panobinostat in patients with castration-resistant prostate cancer. Cancer Chemother Pharmacol. 2013 Sep;72(3):537-44. doi: 10.1007/s00280-013-2224-8. Epub 2013 Jul 3. PMID 23820963

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 35 participants were enrolled in the study at 8 centers in 2 countries- Canada (3 sites) and the United states (5 sites) from 18 March 2008 to 05 November 2010.
Period: Overall Study
Arm/Group | Panobinostat
Started | 35
Completed (Completed here refers to participants who completed study treatment.) | 0
Not Completed | 35
Not completed — Adverse Event | 9
Not completed — Death | 1
Not completed — Disease Progression | 22
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis set (FAS) population included all participants who received at least 1 dose of study drug.
Groups:
- Panobinostat: Participants with metastatic hormone refractory prostate cancer received 20 mg/m^2 of panobinostat i.v. on Days 1 and 8 of a 21-day cycle. Treatment continued until disease progression as per investigator, intolerable toxicity, start of new cancer therapy, death, or withdrawal of consent.
Arm/Group | Panobinostat
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (9.41)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression-Free Survival (PFS) Rate at 24 Weeks
Description: The PFS rate was defined as the percentage of participants that were alive without documented disease progression at the end of 24 weeks from first study treatment. Disease Progression as per response evaluation criteria in solid tumors (RECIST) criteria: Measurable lesions: If target lesion was lymph node then it had to be at least 2 centimeter (cm) at baseline to assess change in size. Bone lesions: (non-target lesions) appearance of greater than or equal to (>=) 2 unequivocal new lesions confirmed on a second scan at least 6 weeks later.
Time Frame: 24 weeks
Population: FAS population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Panobinostat
Number analyzed (Participants) | 35
percentage of participants | 11.4

2. Secondary Outcome: Percentage of Participants With Tumor Response Rate
Description: The tumor response rate was defined as a percentage of participants with confirmed Complete Response (CR) or Partial Response (PR) per RECIST criteria. CR: Disappearance of all target lesions and all nontarget lesions. PR: At least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters.
Time Frame: Every 12 weeks up to approximately 2.7 years
Population: FAS population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Panobinostat
Number analyzed (Participants) | 35
percentage of participants | 0

3. Secondary Outcome: Percentage of Participants With Duration of Stable Disease (SD) Per RECIST
Description: Duration of SD was the time from date of start of treatment to the date of event, defined as the first documented disease progression or death due to underlying cancer. Disease Progression as per RECIST criteria: Measurable lesions: If target lesion was lymph node then it had to be at least 2 cm at baseline to assess change in size. Bone lesions: (non-target lesions) appearance of >=2 unequivocal new lesions confirmed on a second scan at least 6 weeks later. SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD. CR: Disappearance of all target lesions and all nontarget lesions. PR: At least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters. If a participant had not had an event, duration of SD was to be censored at the date of last assessment.
Time Frame: Every 12 weeks up to approximately 2.7 years
Population: We have exhausted all efforts to locate this data and it has since been destroyed, therefore no data is available to report for this outcome measure.
Arm/Group | Panobinostat
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage of Participants With Prostate Specific Antigen (PSA) Response Rate at 24 Weeks
Description: The PSA response was defined as a 50% decrease in PSA from baseline maintained for >= 4 weeks, and without clinical or radiographic evidence of disease progression during this time period. Disease Progression as per RECIST criteria: Measurable lesions: If target lesion was lymph node then it had to be at least 2 cm at baseline to assess change in size. Bone lesions: (non-target lesions) appearance of >= 2 unequivocal new lesions confirmed on a second scan at least 6 weeks later.
Time Frame: 24 weeks
Population: FAS population included all participants who received at least 1 dose of study drug. Overall number of participants analyzed signifies the number of participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Panobinostat
Number analyzed (Participants) | 34
percentage of participants | 0

5. Secondary Outcome: Percentage of Participants With PSA Progression Rate at 24 Weeks
Description: The PSA progression was defined as a 50% rise from nadir and a minimum rise of 2 nanogram per milligram (ng/mL). Disease Progression as per RECIST criteria: Measurable lesions: If target lesion was lymph node then it had to be at least 2 cm at baseline to assess change in size. Bone lesions: (non-target lesions) appearance of >=2 unequivocal new lesions confirmed on a second scan at least 6 weeks later.
Time Frame: 24 weeks
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Panobinostat
Number analyzed (Participants) | 34
percentage of participants | 48.6

6. Secondary Outcome: Median Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of start of treatment to the date of first documented disease progression or death due to any cause. If a participant had not had a disease progression and was alive, the participant was to be censored using the RECIST. Disease Progression as per RECIST criteria: Measurable lesions: If target lesion was lymph node then it had to be at least 2 cm at baseline to assess change in size. Bone lesions: (non-target lesions) appearance of >=2 unequivocal new lesions confirmed on a second scan at least 6 weeks later. Kaplan-Meier method was to be used to estimate the median PFS.
Time Frame: After every cycle up to approximately 2.7 years
Population: as for outcome 3
Arm/Group | Panobinostat
Number analyzed (Participants) | 0

7. Secondary Outcome: Overall Survival
Description: The overall survival was defined as the time from date of start of treatment to date of death due to any cause. If a participant was not known to have died, survival was to be censored at the date of last contact. Kaplan-Meier method was to be used to estimate overall survival.
Time Frame: Start of study treatment to date of death due to any cause (Up to approximately 2.7 years)
Population: as for outcome 3
Arm/Group | Panobinostat
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was an adverse medical event which occurs in a participant of the study and which is not necessarily in a causal relationship with the treatment the participant receives. SAEs were AEs leading to death, are life-threatening, require hospitalizations or prolongation of hospitalizations, represent an innate malformation or a congenital abnormality.
Time Frame: From start of the study up to at least 4 weeks following the last dose of study treatment (Up to approximately 2.7 years)
Population: Safety set population included all participants who were randomized and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat
Number analyzed (Participants) | 35
Participants
  AEs | 35
  SAEs | 14

ADVERSE EVENTS:
Time Frame: From start of the study up to at least 4 weeks following the last dose of study treatment (Up to approximately 2.7 years)
Description: An AE was an adverse medical event which occurs in a participant of the study and which is not necessarily in a causal relationship with the treatment the participant receives. SAEs were AEs leading to death, are life-threatening, require hospitalizations or prolongation of hospitalizations, represent an innate malformation or a congenital abnormality.
Groups:
- Panobinostat: Participants with metastatic hormone refractory prostate cancer received 20 mg/m^2 of panobinostat intravenously (i.v.) on Days 1 and 8 of a 21-day cycle. Treatment continued until disease progression as per investigator, intolerable toxicity, start of new cancer therapy, death, or withdrawal of consent.
Arm/Group | Panobinostat
All-Cause Mortality (participants affected / at risk) | 1/35
Serious Adverse Events (participants affected / at risk) | 14/35
Other Adverse Events (participants affected / at risk) | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat (N=35)
Anaemia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 2
Sepsis (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Blood creatinine increased (Investigations) | 2
Electrocardiogram QT prolonged (Investigations) | 1
Platelet count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Spinal cord compression (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Anuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 1
Ureteric obstruction (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat (N=35)
Anaemia (Blood and lymphatic system disorders) | 6
Leukocytosis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 4
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 16
Atrial fibrillation (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Conjunctival haemorrhage (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 2
Aphthous stomatitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 12
Dry mouth (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 18
Paraesthesia oral (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 11
Asthenia (General disorders) | 2
Axillary pain (General disorders) | 1
Catheter site pain (General disorders) | 1
Chills (General disorders) | 2
Fatigue (General disorders) | 22
Feeling cold (General disorders) | 1
Gait disturbance (General disorders) | 2
Infusion site extravasation (General disorders) | 1
Non-cardiac chest pain (General disorders) | 3
Oedema peripheral (General disorders) | 4
Pain (General disorders) | 1
Pyrexia (General disorders) | 5
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Food allergy (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Candidiasis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 2
Device related infection (Infections and infestations) | 1
Escherichia infection (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Infected cyst (Infections and infestations) | 2
Lung infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 3
Activated partial thromboplastin time prolonged (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 5
Blood creatine increased (Investigations) | 1
Blood creatinine increased (Investigations) | 3
Blood magnesium decreased (Investigations) | 1
Blood phosphorus decreased (Investigations) | 3
Blood potassium decreased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 2
Electrocardiogram ST segment abnormal (Investigations) | 1
Electrocardiogram T wave inversion (Investigations) | 1
Haemoglobin decreased (Investigations) | 6
High density lipoprotein decreased (Investigations) | 1
International normalised ratio increased (Investigations) | 2
Platelet count decreased (Investigations) | 4
Transaminases increased (Investigations) | 1
Weight decreased (Investigations) | 11
Decreased appetite (Metabolism and nutrition disorders) | 13
Dehydration (Metabolism and nutrition disorders) | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 10
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Post herpetic neuralgia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Nocturia (Renal and urinary disorders) | 1
Urinary hesitation (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 2
Penile discharge (Reproductive system and breast disorders) | 1
Penile haemorrhage (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 5
Orthostatic hypotension (Vascular disorders) | 1
Peripheral coldness (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.